CLINICAL TRIAL: NCT06612385
Title: Significance of Platelet Indices and Ratios in Different Degrees of Burn
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Lubna Mansour Shhat Wahba, principal investigator, Assiut University
Other Study IDs: PltIs and PltR in burn degrees
Record Dates: First submitted 2024-09-09; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Platelet Indices; Platelet Ratios

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: platelet indices — Significance of platelet indices and ratios in different degrees of burn

SUMMARY:
Study the correlation between the platelet indices and different degrees of burn Study the correlation between the platelet ratios and different degrees of burn.

DETAILED DESCRIPTION:
Burns are a major traumatic pathology characterized by tissue destruction and cellular degradation resulted by energy transfer and mainly affect skin, which serve as significant cause of morbidity and mortality. burns are classified as first,second and third degree depending on how deep and severe they penetrate the skin surface.

Platelets play important role in primary homeostasis, thrombosis, inflammation and tissue regulation in the processes of wound healing. Platelets can contact exposed collagen and extra cellular matrix and releasing clotting factors to achieve homeostasis as well as essential growth factors and cytokines to repair the wound.In clinical, Platelet-rich plasma (PRP) is a concentrate of autologous platelets,has been used to effectively accelerate burn wound healing Platelet indices (PI), markers of platelet activation, are parameters obtained daily as a part of an automatic blood count, Platelet indices are related to platelets morphology and proliferation kinetics. Most commonly assessed platelet indices include the mean platelet volume (MPV), mean distribution width(PDW),Platelet larger cell ratio (PLCR) ,platelet crit (PCT), mean platelet mass (MPM),mean platelet component (MPC),Platelet component distribution width (PCDW) and immature platelet fraction (IPF).

The ratio of red blood cell distribution width (RWD) and platelet (PLT) (RPR) is considered an inflammation biomarker associated with the poor prognosis of number of diseases. There is two studies about PRP related to prognosis of major burn injury . results indicate that RPR-as an inflammatory index- can be used as a biomarker for prognosis of adult patients with major burn injuries.

Blood-based platelet parameters, due to their fairly easy accessibility and inexpensive methods of measurement, seem to be on the rise as potential novel biomarkers of numerous ,both acute and chronic disease. However, To date ,there are no data on the significance of platelets indices in evaluation with different degrees of burn .In this study we will evaluate the significance of platelet ratios and indices in different degrees of burn.

ELIGIBILITY:
Inclusion Criteria:

* burn degree ( 1,2,3)

Exclusion Criteria:

* patient with ITB

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study the correlation between the platelet indices and different degrees of burn Study the correlation between the platelet ratios and different degrees of burn.
Sampling Method: Non-Probability Sample
Enrollment: 333 (Estimated)
Dates: Start 2024-10-10 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Significance of platelet indices in different degrees of burn | basline
  Study the correlation between the platelet indices and different degrees of burn
Significance of platelet ratios in different degrees of burn | basline
  Study the correlation between the platelet ratios and different degrees of burn.